CLINICAL TRIAL: NCT06176989
Title: Phase II Study of Enasidenib in IDH2-mutated Malignant Sinonasal and Skull Base Tumors
Brief Title: Enasidenib in IDH2-Mutated Malignant Sinonasal and Skull Base Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001552; 001552-C
Record Dates: First submitted 2023-12-19; First posted 2023-12-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10-16

CONDITIONS: Metastatic Chondrosarcoma; Locally Advanced Chondrosarcoma; Metastatic Sinonasal Adenocarcinoma; Locally Advanced Sinonasal Adenocarcinoma; Metastatic Large-cell Neuroendocrine Carcinoma; Locally Advanced Large-cell Neuroendocrine Carcinoma; Metastatic Olfactory Neuroblastoma; Locally Advanced Olfactory Neuroblastoma; Metastatic Sinonasal Undifferentiated Carcinoma; Locally Advanced Sinonasal Undifferentiated Carcinoma
Keywords: R140 mutation; R172 mutation; Small Molecule Inhibitor
MeSH Terms: conditions — Chondrosarcoma; Esthesioneuroblastoma, Olfactory; Sinonasal undifferentiated carcinoma | interventions — enasidenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Participants with IDH2 mutated (R140/R172) malignant sinonasal and skull base tumors.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — 100mg PO (orally) once daily, on days 1-28 of a 28-day cycle

SUMMARY:
Background:

Cancers of the nasal cavity or skull base are rare. They often are not diagnosed until they are at an advanced stage, and they often spread to other parts of the body. These cancers may have mutations in a gene called IDH2. Researchers want to find out if a drug (enasidenib) that targets the IDH2 mutation can help people with these cancers.

Objective:

To test enasidenib in people with cancers of the nasal cavity or skull base.

Eligibility:

People aged 18 years and older with rare cancers of the nasal cavity or the base of the skull. Their cancer must have an IDH2 gene mutation, and it must have recurred locally or spread to other parts of the body. These cancers can include sinonasal undifferentiated carcinoma; olfactory neuroblastoma; sinonasal large-cell neuroendocrine carcinoma; poorly differentiated sinonasal adenocarcinoma; or chondrosarcoma.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests and tests of their heart function. They will have imaging scans of their brain, skull base, neck, chest, abdomen, and pelvis. A sample of tumor tissue will be collected.

Enasidenib is a tablet taken by mouth with a glass of water. Participants will take the drug once a day, every day, in 28-day cycles. They will not have resting periods between cycles.

Participants will visit the clinic on the first day of each cycle to receive the tablets they will need to take at home until the beginning of the next cycle. They will keep a diary to record the time of each dose they take.

Participants may remain in the study as long as the drug is helping them....

DETAILED DESCRIPTION:
Background:

* Sinonasal undifferentiated carcinoma (SNUC) and olfactory neuroblastoma (ONB) are rare malignant sinonasal and skull base tumors, a group that also includes sinonasal adenocarcinoma, squamous cell carcinoma, large cell neuroendocrine carcinoma, sinonasal papilloma, chondrosarcoma (CS), chordoma and others.
* These malignancies are often diagnosed at a locally advanced stage. They tend to invade locally and have high rates of regional spread to the neck, and distally to the lungs and bones. For early locoregional disease multimodality treatment is used: surgery with postoperative radiotherapy, with or without induction chemotherapy. Treatment approaches for metastatic disease are largely based on institutional case series and consist largely of systemic chemotherapy.
* Recent genomic studies have reported isocitrate dehydrogenase-2 (IDH2) hotspot mutations in up to 87% of SNUC, 17% of ONB, and in 12% of chondrosarcomas; it has also been reported in sinonasal large-cell neuroendocrine carcinoma (LCNEC) and poorly differentiated sinonasal adenocarcinoma (SNAC).
* IDH2 hotspot mutations have been identified in acute myeloid leukemia, glioblastoma, myelodysplastic syndromes, and cholangiocarcinoma.
* Enasidenib is an orally bioavailable, selective and potent inhibitor of mutated IDH2, which is approved in relapsed IDH2 mutated (IDH2m) AML.
* Inhibition of mutated IDH2 may be clinically useful in IDH2m malignant sinonasal and skull base tumors.

Objectives:

- To estimate the overall progression free survival (PFS) based on treatment with enasidenib in all study participants with IDH2m malignant sinonasal and skull base tumors.

Eligibility:

* Histologically or cytologically confirmed locally advanced or metastatic SNUC, ONB, LCNEC, SNAC, and CS with documented somatic (tumor) IDH2 mutations R140 or R172.

  * Eligible primary tumor locations are sinonasal cavity and skull base.
  * Locally advanced disease must not be amenable to potentially curative surgery/radiotherapy.
  * Must have recurred or progressed following prior systemic therapy administered in the recurrent or metastatic setting. Any number of prior systemic therapies is allowed
* Measurable disease, per RECIST 1.1
* Age >= 18 years
* ECOG Performance Status 0-2
* Adequate organ function

Design:

* Single-arm Phase II trial to determine PFS in participants with recurrent or metastatic IDH2m malignant sinonasal and skull base tumors.
* Enasidenib will be given at a dose of 100mg orally once daily until progressive disease or unacceptable toxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed locally advanced or metastatic SNUC, ONB, LCNEC, SNAC, and CS with documented somatic (tumor) IDH2 mutations R140 or R172. Primary tumors must be located in the sinonasal cavity and/or skull base.
* Locally advanced disease must not be amenable to potentially curative surgery/radiotherapy.
* Must have recurred or progressed following prior systemic therapy administered in the recurrent or metastatic setting. Any number of prior systemic therapies is allowed.
* Measurable disease, per RECIST 1.1. Lesions in a previously irradiated field are considered measurable if they have been demonstrated as progressing during or following radiotherapy.
* Age >=18 years.
* ECOG performance status 0-2
* Adequate organ and marrow function as defined below:

  * hemoglobin >=9 g/dL (PRBC transfusion allowed)
  * absolute neutrophil count (ANC) >=1,000/mcL
  * platelets >=75,000/mcL
  * total bilirubin <= 1.5 x institutional upper limit of normal (iULN) (<=3x in the presence of Gilbert s syndrome or a UGT1A1 gene mutation)
  * AST/ALT <=1.5 x iULN (<=2.5 x iULN if liver metastasis)
  * Serum Creatinine <=1.5 x iULN OR
  * Creatinine Clearance >=40 mL/min by Cockroft-Gault GFR estimation for subjects with serum creatinine levels <=1.5 X iULN
* Participants with treated brain or central nervous system metastases are eligible if follow-up brain imaging after at least 4 weeks following CNS-directed therapy shows no evidence of progression.
* Participants positive for human immunodeficiency virus (HIV) must have CD4 count >= 200 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy for at least 4 weeks and have no reported opportunistic infections or Castleman s disease within 12 months prior to treatment.
* Participants with evidence of chronic hepatitis B virus (HBV) infection, must have HBV viral load that is undetectable on suppressive therapy, if indicated.
* Participants with evidence of HCV infection, must have viral load that is undetectable.
* Women of reproductive potential (WORP*) and men with female partners of reproductive potential must agree to abstain from sexual intercourse or to use 1 highly effective method of contraception during the study and for at least 2 months following the last dose of enasidenib. A highly effective form of contraception is one of the following: hormonal contraception (e.g., oral contraceptive pills, intravaginal ring, transdermal patch, injection, implant); intrauterine device (IUD); tubal ligation; or a partner with a vasectomy.
* Participants who are breastfeeding or plan to breastfeed must agree to discontinue/postpone breastfeeding while on study therapy and for at least 2 months after the last dose.
* Ability of participant to understand and willingness to sign a written informed consent document.
* Willingness to provide blood samples and undergo biopsy of tumor for research purposes. Participants may be exempt from biopsy.
* Participants must co-enroll in companion protocol study #18-DC-0051 entitled Biospecimen procurement for NIDCD clinical protocols . A separate informed consent will be obtained from study participants for this study.
* Participants with ONB must co-enroll in companion protocol #21-C-0009 entitled A Natural History Study of Children and Adults with Olfactory Neuroblastoma . A separate informed consent will be obtained from study participants for this study.

  * WORP: any woman who has experienced menarche and has not had hysterectomy or bilateral oophorectomy or is not postmenopausal (amenorrheic 12 months or more following cessation of exogenous hormonal treatments; if <50 years old need follicle stimulating hormone FSH in the post-menopausal range)

EXCLUSION CRITERIA:

* Prior treatment with IDH1/2 inhibitor.
* Use of other investigational agents within 3 weeks or 5 half-lives prior to first treatment administration.
* Systemic anticancer treatment within 3 weeks prior to first treatment administration. All residual treatment-related toxicities must have resolved or be minimal and not constitute a safety risk. Note: Bisphosphonates and denosumab are permitted medications.
* Large-field radiotherapy within 4 weeks prior to first treatment administration. All residual treatment-related toxicities must have resolved (except xerostomia) or be minimal and not constitute a safety risk.
* Major surgery within 2 weeks prior to first treatment administration. If participant underwent major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. Minimally invasive procedures are permitted.
* Participants with new or progressive (active) brain metastases or leptomeningeal disease.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enasidenib.
* Treatment with botanical preparations (e.g., herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to first treatment administration.
* Participants taking the following sensitive cytochrome P450 (CYP) substrate medications that have a narrow therapeutic range are excluded from the study unless they can be transferred to other medications prior to enrolling: warfarin, phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline and tizanidine (CYP1A2). Excluded medications should not be given within 3 weeks or 5 half-lives (whichever is shorter) prior to the first dose of study medication. Other CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP1A2 substrates may be given concurrently if medically necessary.
* Participants taking sensitive substrates of P-glycoprotein (P-gp), breast cancer resistant protein (BCRP), OAT1, OATP1B1, OATP1B3, and OCT2 should be excluded from the study unless the substrate medication can be dose modified according to the package insert of the substrate (if applicable) and adverse events can be closely monitored during concurrent administration. Alternately, participants can be transferred to other medications prior to enrolling. Excluded medications should not be given within 3 weeks or 5 half-lives (whichever is shorter) prior to the first of study medication.
* Participants taking medications that are known to prolong the QT interval unless the participant can be transferred to other medications at least 5 half-lives prior to the start of the study treatment. If equivalent medication is not available, QTc will be closely monitored
* Impaired cardiovascular function or clinically significant cardiovascular disease, including, but not limited to, any of the following:

  * cerebral vascular accident/stroke (< 3 months prior to enrollment),
  * uncontrolled hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >100 mmHg)
  * acute coronary syndromes (including myocardial infarction < 6 months prior to enrollment, unstable angina),
  * Symptomatic congestive heart failure
  * Rate-corrected QT (QTc using Fridericia formula [QTcF]) >450 msec
  * Severe/uncontrolled ventricular arrhythmia
* Known short-gut syndrome, gastroparesis, or other conditions that limit the ingestion of gastrointestinal absorption of drugs administered orally.
* Active infection requiring treatment with parenteral antibiotics.
* History of second malignancy within 3 years prior to enrollment except for the following: adequately treated localized basal cell or squamous skin cancer, cervical carcinoma in situ, superficial bladder cancer, other localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk CLL).
* Participant pregnancy
* Uncontrolled intercurrent illness (including psychiatric) or social situations, that may limit interpretation of results or increase risk to the participant:

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in all study participants | up to 5 years post study treatment
  The date of first treatment until the date of disease progression or death without progression

SECONDARY OUTCOMES:
safety | from study treatment initiation up to 28 days post study treatment
  Adverse events assessed per CTCAE version 5
clinical benefit rate (CBR: CR+PR+SD>4 months) in participants with IDH2m SNUC | up to 5 years post study treatment
  Fraction of participants experiencing CBR = CR+PR+ SD > 16 weeks
PFS in non-SNUC IDH2m tumors | up to 5 years post study treatment
  The date of first treatment until the date of disease progression or death without progression
Overall survival (OS) in non-SNUC IDH2m tumors | up to 5 years post study treatment
  The date of first treatment until date of death or last follow-up
clinical benefit rate (CBR: CR+PR+SD>4 months) in participants with non-SNUC IDH2m tumors | up to 5 years post study treatment
  Fraction of participants experiencing CBR = CR+PR+ SD > 16 weeks
Overall survival (OS) in participants with IDH2m SNUC | up to 5 years post study treatment
  The date of first treatment until date of death or last follow-up
PFS in participants with IDH2m SNUC | up to 5 years post study treatment
  The date of first treatment until the date of disease progression or death without progression
Correlate UGTIA1 genotypes with toxicity | from study treatment initiation up to 28 days post study treatment
  Descriptive statistics of AE occurence per UGTIA1 genotype

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.@@@@@@
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing. This study will comply with the NIH Genomic Data Sharing (GDS) Policy, which applies to all new and ongoing NIH IRP-funded research, as of January 25, 2015, that generates large-scale human or non-human genomic data, as well as the use of these data for subsequent research. Large-scale data include genome-wide association studies (GWAS), single nucleotide polymorphisms (SNP) arrays, and genome sequence, transcriptomic, epigenomic, and gene expression data. Therefore, unlinked genomic data will be deposited in public genomic databases such as dbGaP in compliance with the NIH Genomic Data Sharing Policy.@@@@@@@@@@@@
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.@@@@@@

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001552-C.html